CLINICAL TRIAL: NCT02700828
Title: Prospective, Randomized, Double-blind, Cohort Study of Hydrocortisone vs Placebo in Systemic Low Blood Pressure During Hypothermia Treatment in Asphyxiated Newborns
Brief Title: Hydrocortisone Treatment In Systemic Low Blood Pressure During Hypothermia in Asphyxiated Newborns
Acronym: CORTISoL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Agnes Jermendy MD PhD MPH, assistant lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1Ped-AsphCort 001
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Asphyxia
Keywords: Hypothermia treatment; Circulatory failure; Neonatal hypotension; Relative adrenal insufficiency; Hydrocortisone supplementation
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia; Shock | interventions — Hydrocortisone; hydrocortisone hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone (Active Comparator): Hydrocortisone is the pharmaceutical term for cortisol, the principal glucocorticoid secreted by the adrenal gland
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Isotonic sodium chloride is an aqueous solution of 0.9 percent sodium chloride which is isotonic with the blood and tissue fluid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — 4 * 0,5 mg/kg /24 hours (in every 6 hours) iv., during hypothermia treatment (max. 72 hours)
  Other Names: Solu-Cortef
  Arms: Hydrocortisone
Drug: Placebo — 4 * 2 ml isotonic sodium chloride solution /24 hours (in every 6 hours) iv., during hypothermia treatment (max. 72 hours)
  Other Names: Isotonic saline
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo controlled, single center study to compare low dose hydrocortisone vs placebo in systemic low blood pressure during hypothermia treatment in asphyxiated newborns. Patients will be allocated to one of the treatment arms (hydrocortisone or placebo) while receiving conventional inotropic therapy as needed.

The hypothesis is that cooled asphyxiated neonates develop relative adrenal insufficiency that may contribute to hypotension and lower efficacy of inotropic therapy in this patient population. Thus, the investigators are planning to measure initial serum cortisol levels and investigate the cardiovascular effects of low dose hydrocortisone supplementation besides conventional inotropic therapy in a placebo-controlled fashion.

DETAILED DESCRIPTION:
Hypothesis:

The researchers hypothesized that asphyxiated neonates undergoing therapeutic hypothermia develop relative adrenal insufficiency that contributes to "late onset" (>24 hours after birth) hypotension resistant to optimized pharmacological support.

Thus, the investigators are planning to measure initial serum cortisol levels and investigate the cardiovascular effects of low dose hydrocortisone supplementation.

Specific aims:

1. To study initial serum cortisol levels in asphyxiated newborns undergoing therapeutic hypothermia with late onset hypotension.
2. To demonstrate that in asphyxiated newborns undergoing therapeutic hypothermia and presenting with systemic hypotension resistant to optimized pharmacological support, low dose hydrocortisone supplementation restores normal blood pressure when compared to placebo.

Methodology:

* Prospective, randomized, double-blind, single center, cohort study
* 1st Department of Paediatrics, NICU, Semmelweis University, Hungary
* Starting date: 02/14/2016
* Patient number: 16 vs 16 (hydrocortisone vs placebo - based on previous observational study results)
* Intervention (hydrocortisone vs placebo) applied only during therapeutic hypothermia (max. 72 hours)
* Neurodevelopmental follow-up visit: Bayley II/III scale to evaluate the effect of hydrocortisone treatment on the neurological development at the age between 18 and 22 months.

Drugs for hypotension, the hydrocortisone protocol:

1. Fluid replacement (volume bolus: 10-20 ml/kg isotonic saline, over 15 minutes, according to the clinician's decision)
2. In case of persisting hypotension: serum sample is collected for cortisol measurement.
3. Randomization, irrespective of actual cortisol level. As the study is blinded, enrollment in the clinical trial will/shall not influence the clinical decision making about further interventions. A dedicated study assistant will be available to prepare the drug / placebo for the newborns.

   * Inotropic therapy (dopamine, following the standard titration protocol)
   * AND (at start of dopamine) hydrocortisone: 4 * 0,5 mg/kg /24 hours (in every 6 hours) or placebo administration (the corresponding amount of isotonic saline)
4. After randomization, intervention is continued until the end of hypothermia treatment (max. 72 hours), with the same dose. Inotropic therapy will be titrated as needed.

ELIGIBILITY:
Inclusion Criteria:

1. The infant will be assessed sequentially by criteria A, B and C, as described by the TOBY trial and listed below, to be eligible for hypothermia treatment.

   A. Infants ≥ 36 completed weeks of gestation admitted to the NICU with at least one of the following:
   * Apgar score of ≤ 5 at 10 minutes after birth
   * Continued need for resuscitation, including endotracheal or mask ventilation, at 10 minutes after birth
   * Acidosis within 60 minutes of birth (defined as any occurrence of umbilical cord, arterial or capillary pH < 7.00)
   * Base Deficit ≥ 16 mmol/L in umbilical cord or any blood sample (arterial, venous or capillary) within 60 minutes of birth

   B. Moderate to severe encephalopathy, consisting of altered state of consciousness (lethargy, stupor or coma) AND at least one of the following:
   * hypotonia
   * abnormal reflexes including oculomotor or pupillary abnormalities
   * absent or weak suck
   * clinical seizures

   C. At least 30 minutes duration of aEEG recording that shows abnormal background aEEG activity or seizures. There must be one of the following:
   * normal background with some seizure activity
   * moderately abnormal activity
   * suppressed activity
   * continuous seizure activity
2. Invasive arterial blood pressure measurement: umbilical arterial catheter or peripheral arterial catheter to measure invasively the arterial blood pressure.
3. During hypothermia treatment low blood pressure was detected and treated with the following:

   * fluid therapy: 10-20 ml/kg isotonic NaCl if hypotension is still present
   * inotropic therapy: dopamine in parallel with study intervention
4. A written informed consent has been obtained from a parent of each infant after explanation of the study.

Exclusion Criteria:

1. Signed informed consent is unavailable.
2. Infants who are expected to be > 6 hours of age (not suitable for cooling).
3. Congenital abnormalities, cardiac anomalies, meconium aspiration syndrome.
4. Low blood pressure coincides with high heart rate (>120/min) in cooled infants, suggesting hypovolaemia.
5. Haematocrit level < 35%.
6. Need for combined, ≥2 types of inotropic therapy.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Compare mean arterial blood pressure (MAP) change in the patients receiving hydrocortisone vs placebo | 2 hours
  Circulatory stability as measured by an increased MAP (5 mmHg) within two hours after drug administration

SECONDARY OUTCOMES:
Frequency of initially low serum cortisol in hypotensive asphyxiated newborns undergoing therapeutic hypothermia | before hydrocortisone administration within max. 72 hours
  Initially low serum cortisol - proven relative adrenal insufficiency
Length of dopamine treatment in the patients receiving hydrocortisone vs placebo | 72 hours
  Compare dopamine treatment's length (in hours) in the patients receiving hydrocortisone vs placebo
Cumulative dopamine dose in the patients receiving hydrocortisone vs placebo | 72 hours
  Compare cumulative dopamine dose (mcg/kg) in the patients receiving hydrocortisone vs placebo
Change in hourly diuresis in the patients receiving hydrocortisone vs placebo | 72 hours
  Measure and compare the hourly diuresis (ml/kg/hour) in the patients receiving hydrocortisone vs placebo
Change in the echocardiography parameters (fractional shortening and cardiac output) in the patients receiving hydrocortisone vs placebo | 72 hours
  Fractional shortening (FS%) and cardiac output (CO in ml/kg/min) measurements before and after hydrocortisone or placebo, during the first 72 hours (during hypothermia treatment)
Long term neurodevelopmental outcome in the patients receiving hydrocortisone vs placebo | 18-22 month
  Performance on motor and mental scales of Bayley II/III scales of infant development

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Szabó, MD, PhD, Study Director — Semmelweis University, 1st Department of Paediatrics
Locations (1):
- Semmelweis University, 1st Department of Paediatrics, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Noori S, Friedlich P, Wong P, Ebrahimi M, Siassi B, Seri I. Hemodynamic changes after low-dosage hydrocortisone administration in vasopressor-treated preterm and term neonates. Pediatrics. 2006 Oct;118(4):1456-66. doi: 10.1542/peds.2006-0661. PMID 17015536
- [Background] Ibrahim H, Sinha IP, Subhedar NV. Corticosteroids for treating hypotension in preterm infants. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003662. doi: 10.1002/14651858.CD003662.pub4. PMID 22161379
- [Background] Rios DR, Moffett BS, Kaiser JR. Trends in pharmacotherapy for neonatal hypotension. J Pediatr. 2014 Oct;165(4):697-701.e1. doi: 10.1016/j.jpeds.2014.06.009. Epub 2014 Jul 16. PMID 25039051
- [Background] Hebbar KB, Stockwell JA, Leong T, Fortenberry JD. Incidence of adrenal insufficiency and impact of corticosteroid supplementation in critically ill children with systemic inflammatory syndrome and vasopressor-dependent shock. Crit Care Med. 2011 May;39(5):1145-50. doi: 10.1097/CCM.0b013e31820eb4e4. PMID 21336126
- [Background] Ng PC, Lam CW, Fok TF, Lee CH, Ma KC, Chan IH, Wong E. Refractory hypotension in preterm infants with adrenocortical insufficiency. Arch Dis Child Fetal Neonatal Ed. 2001 Mar;84(2):F122-4. doi: 10.1136/fn.84.2.f122. PMID 11207229
- [Background] Ng PC, Lee CH, Bnur FL, Chan IH, Lee AW, Wong E, Chan HB, Lam CW, Lee BS, Fok TF. A double-blind, randomized, controlled study of a "stress dose" of hydrocortisone for rescue treatment of refractory hypotension in preterm infants. Pediatrics. 2006 Feb;117(2):367-75. doi: 10.1542/peds.2005-0869. PMID 16452355
- [Background] Seri I, Tan R, Evans J. Cardiovascular effects of hydrocortisone in preterm infants with pressor-resistant hypotension. Pediatrics. 2001 May;107(5):1070-4. doi: 10.1542/peds.107.5.1070. PMID 11331688
- [Result] Kovacs K, Szakmar E, Meder U, Szakacs L, Cseko A, Vatai B, Szabo AJ, McNamara PJ, Szabo M, Jermendy A. A Randomized Controlled Study of Low-Dose Hydrocortisone Versus Placebo in Dopamine-Treated Hypotensive Neonates Undergoing Hypothermia Treatment for Hypoxic-Ischemic Encephalopathy. J Pediatr. 2019 Aug;211:13-19.e3. doi: 10.1016/j.jpeds.2019.04.008. Epub 2019 May 30. PMID 31155392
- [Derived] Kovacs K, Szakmar E, Dobi M, Varga Z, Meder U, Szabo AJ, McNamara PJ, Szabo M, Jermendy A. Neurodevelopmental outcome in infants with neonatal encephalopathy receiving hydrocortisone during therapeutic hypothermia: follow-up of the extended-CORTISoL trial. J Perinatol. 2025 Dec;45(12):1788-1794. doi: 10.1038/s41372-025-02428-5. Epub 2025 Sep 22. PMID 40983658